CLINICAL TRIAL: NCT02170337
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 282 in Healthy Subjects and Subjects With Chronic Rhinosinusitis With Nasal Polyps
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 282 in Healthy Subjects and Subjects With Chronic Rhinosinusitis With Nasal Polyps
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110236
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 282 (Experimental): AMG 282 administered as subcutaneous and intravenous doses.
  Interventions: Drug: AMG 282
- Placebo (Placebo Comparator): No active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 282 — AMG 282 is for the treatment of subjects with chronic rhinosinusitis with nasal polyps
  Arms: AMG 282
Drug: Placebo — Contains no active drug
  Arms: Placebo

SUMMARY:
A randomized, double-blind, ascending multiple dose study in healthy volunteers and subjects with chronic rhinosinusitis with nasal polyps

ELIGIBILITY:
Healthy Volunteers:

Inclusion Criteria:

* Healthy males and females witha BMI between 18.0 and 32.0 kg/m2, inclusive

Exclusion Criteria:

* subject with evidence of a clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with study evaluation, procedures, or completion.

Subjects with chronic rhinosinusitis with nasal polyps (CRSwNP):

Inclusion Criteria:

* diagnosis of CRSwNP (inflammation of the nose and paranasal sinuses characterized in adults by 2 or more symptoms, 1 of which should be either nasal blockage or nasal discharge and/or facial pain and/or reduced smell for greater than 12 weeks)
* bilateral nasal polyps of grade 3 or 4

Exclusion Criteria:

* Forced Expiratory Volume (FEV1) </= 70%
* Asthma exacerbation requiring systemic corticosteroid treatment or hospitalization for > 24h for treatment of asthma, within 3 months prior to screening or are on a dose of greater than 1000 μg fluticasone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 169 days
  Subject incidence of treatment-emergent adverse events, vital signs, physical examinations, laboratory safety tests, and 12-lead electrocardiograms (ECGs)
Immunogenicity | 169 days
  Subject incidence of anti-AMG 282 antibodies

SECONDARY OUTCOMES:
Pharmacokinetic profile of AMG 282 | 169 days
  Serum concentrations and derived PK parameters (eg, time to maximum concentration [tmax], area under the concentration-time curve over the dosing interval τ [AUCτ] after the first and last dose, and maximum observed concentration [Cmax]).

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - Research Site, Santa Monica, California
  - Research Site, Aurora, Colorado
  - Research Site, South Miami, Florida
  - Research Site, Houston, Texas

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com